CLINICAL TRIAL: NCT03051763
Title: PEGASUS - The Effects of Commercial Air Travel on Patients Suffering From Pulmonary Hypertension: A Prospective, Multicentric Analysis
Brief Title: The Effects of Commercial Air Travel on Patients Suffering From Pulmonary Hypertension
Acronym: PEGASUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); DRK Kliniken Berlin Köpenick, Berlin, Germany (Unknown); University Hospital, Zürich (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Principal Investigator, Jan Grimminger, MD, University of Giessen
Other Study IDs: 204/16
Record Dates: First submitted 2017-02-01; First posted 2017-02-14 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; commercial air travel
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to 1) descriptively report possible in flight events and 2) to provide regression analysis if the number of events are statistically significant in their prevalence and thus are useful in finding possible parameters in echocardiography, right heart catheterization, laboratory findings, spiroergometry as well as six minute walk test to produce a risk assessment for possible expected in flight adverse events as well as a recommendation concerning the need of supplemental oxygen for each individual patient.

The investigators therefore want to find out:

1. In which subgroup (if applicable) of PH patients in flight adverse events are more frequent.
2. Whether there are parameters (from blood samples, blood gas analysis, World Health Organization-Functional Class (WHO-FC), Six Minute Walk (SMW), echocardiography, right heart catheter (RHC)) that are able to predict in flight need for additional oxygen and/or possible adverse events.

DETAILED DESCRIPTION:
Pulmonary Hypertension (PH) is a progressive disease affecting the pulmonary vessels and leading to an increased pulmonary vascular resistance (PVR) and thus right heart strain. The result is an increase in mean pulmonary arterial pressure (mPAP) and with time dilation of the right heart chambers as well as hypertrophy of the right ventricular myocardium. As the increase in PVR progresses further, the right ventricle struggles to cope with the rising afterload and starts to fail. Before this worst case scenario occurs, most individuals suffering from PH notice dyspnea on exertion as the first sign of their underlying disease. The increased proliferation and the resulting rise in PVR lead to a slower blood flow through the pulmonary vessels and thus sometimes result in in situ thrombosis. Furthermore the thickening of the capillary vessel bed increases the diffusion barrier for oxygen and herby results ventilation-perfusion mismatch and leads to hypoxia first during exercise, and later even at rest, making long term oxygen therapy (LTOT) necessary. Today's specific pulmonary-vasoactive therapy helps individuals suffering from PH to live a "normal" life. For most people this also means going on vacation - if necessary by plane. The latter however bares risks for patients suffering from PH:

While the average traveling altitude of passenger planes is between 9.150 - 12.200m (30.000 - 40.000ft) where the atmospheric pressure is less than 30% compared to that at sea level, reducing the pressure of inspired oxygen (PIO2) from 143mmHg to less than 40mmHg. In other words the air contains less than 6% oxygen compared to 21% at sea level. Since this is not compatible with human life airplane cabins are pressurized to maintain a pressure equally to a height between 1520 - 2440m (5.000 - 8.000ft) which contains about 15% of oxygen. However, even the National Research Council (NRC) stated that passengers with cardiovascular problems might experience discomfort within this cabin environment. These conditions of hypobaric hypoxia, even in the pulmonary vasculature of a healthy individual, lead to a generalized hypoxic pulmonary vasoconstriction (HPV). These changes, in healthy individual lead to a rise in PVR and thus right ventricular systolic pressure (RVSP). Healthy individuals are able to compensate the resulting increase in right ventricular afterload. It however is easily imaginable that the heart of a patient with right heart insufficiency may struggle or even fail under these circumstances. Increasing the PIO2 through supplemental oxygen (O2) is known to prevent these changes, which is why it is recommended to be used by patients with world health organization functional class (WHO-FC) III and IV as well as patients with arterial blood O2 pressure consistently <, 60mmHg (8 kPa) by the current guidelines. This general advice is given by the American Aerospace Medical Association and the British Thoracic Society as well. There is however a problem with most of these recommendations: There's a lack of studies concerning the effects of commercial air travel on patients with PH, which is why many recommendations are made by transferring data from surveys about more common lung diseases. There are however some studies on the effects of (simulated) air travel in patients with PH:

In 2012 a survey was conducted where hypoxic challenge test (HCT) was performed on 36 individuals suffering from PH and compared the acquired data of HCT and WHO-FC with the actual need of in flight oxygen. The latter information was gained through a questionnaire handed out to the before named individuals that focused on in flight symptoms and events that lead to the use of in flight oxygen prior to and after diagnosis of PH. It was found that 25 out of the examined 36 individuals according to the current recommendations would need in flight oxygen judging by their WHO-FC, but only 10 failed HCT. Out of all 36 patients, 14 traveled by plane after being diagnosed with PH. Of these, nine subjects should have had in-flight oxygen based on WHO-FC but were asymptomatic without. Furthermore 1 individual that passed the HCT had developed symptoms during the flight and 3 who failed the HCT were asymptomatic flying without oxygen. In other words: HCT did not identify one patient who developed symptoms during a flight.

In the same year another study was published with data of a prospective survey from 34 individuals of which data was collected during flight. Cabin pressure, peripheral oxygen saturation (SpO2), heart rate and symptoms were assessed. Desaturation was defined as SpO2 < 85%. It was found that nine individuals experienced significant desaturation. Furthermore only five out of the 13 patients that reported symptoms presented desaturation during their flight. Furthermore no predictive factor to predict possible desaturation during the time being airborne (neither resting SpO2 at sea level nor maximal estimated cabin altitude was predictive) were found.

In 2011 a retrospective analysis during which patients with diagnosed PH, who had traveled by airplane, were asked to complete a questionnaire containing general information (group of PH, WHO-FC, current medication, usage of LTOT, etc.) as well as possible symptoms conceived (dyspnea, chest pain, peripheral edema, etc.) was released. Out of 179 patients who had traveled by plane 57 were under LTOT and 29 used supplemental oxygen during the flight. In total 20 adverse events were reported (mainly mild to moderate in severity) and 7 needed medical assistance. In total 159 out of 179 patients didn't experience any discomfort during or shortly after their travel.

In summary of the scarce data available hitherto there is no sufficient test available to predict in flight complications in patients with pulmonary hypertension. It could however be shown that using WHO-FC as the only surrogate is not useful to determine which patient might be in need of additional oxygen during air travel. Furthermore even HCT is not capable of detecting patients at risk. Even the British Thoracic Society marks their recommendations on the use of supplemental oxygen for patients with PH with "evidence level D".

It is this absence of sufficient data and the thereby resulting uncertainty of patients, physicians, pneumologist and cardiologists as well as specialists in the field of PH on this topic that lead to the concept of this study. By this prospective survey on patients suffering from all forms of PH, under all different types of available treatments and in all WHO-FCs the investigators hope to gain further insight in possible markers to predict in flight adverse events and thus make flying safer for individuals struggling with PH. This study therefore aims to include a total of 1000 patients suffering from all forms of PH which, after providing written and informed consent, will be asked to fill out a questionnaire prior to and after air traveling as well as assessing vital parameters (SpO2, pulse and respiration rate) prior to, during and shortly after their flight. In addition all clinical data available will be collected and analyzed. The aim of this study is to find possible parameters in echocardiography, right heart catheterization, laboratory findings, spiroergometry as well as six minute walk test to produce a risk assessment for possible expected in flight adverse events as well as a recommendation concerning the need of supplemental oxygen for each individual patient.

All data collected will be anonymised to prevent possible identification of each participating individual. Examinations conducted during this survey would have been necessary anyway in the course of regular clinical visits. So there will be no additional health risk for patients participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* written an informed consent
* invasively diagnosed pulmonary hypertension
* mPAP > 25mmHg
* PAWP < 15mmHg
* PVR < 3WU

Exclusion Criteria:

* missing written and informed consent
* cystic fibrosis
* significant left cardiac impairment
* LVEF < 45%
* history of atrial flutter
* aortic / mitral valve vitium > mild
* history of myocardial infarction
* coronary bypass
* clinically significant anemia (Hb < 8,0g/l).
* malignoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary (arterial) hypertension planing commercial air travel.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-12-19 (Estimated); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 2 years
  Self report of possible (serious) adverse events (desaturation, palpitations, thoracic tightness / pain, dizziness, syncope) during flight by a specific questionnaire. Each symptom may be marked with 1 (occurred) and 0 (did not occur).

SECONDARY OUTCOMES:
Defining possible predictive parameters for patient in flight safety | 2 years
  Reported in flight events will lead to further investigations concerning clinically gained data to find possible markers that are useful in predicting which individual is safe to fly, which should not fly at all and which is recommended to use additional oxygen during the flight.
Defining possible predictive parameters for patient in flight safety in echocardiography | 2 years
  Assessment of TAPSE in mm as well as Tei-Index
Defining possible predictive parameters for patient in flight safety in hemodynamics | 2 years
  Assessment of mPAP in mmHg, PVR in WU as well as CI in l/min/m2
Defining possible predictive parameters for patient in flight safety in spiroergometry | 2 years
  Assessment of VO2max in ml/kg*min
Defining possible predictive parameters for patient in flight safety in six minute walk test | 2 years
  Assessment of covered distance in m, possible desaturation in %, possible changes in blood pressure in mmHg as well as changes in puls in beats/min

CONTACTS AND LOCATIONS:
Overall Officials: Ghofrani H. Ardeschir, Prof. Dr., Study Chair — University of Giessen
Locations (5):
- Germany (4):
  - University Clinic Giessen and Marburg, Giessen, Hesse
  - University Clinic Dresden, Dresden, Saxony
  - DRK Kliniken Berlin, Berlin
  - University Clinic Hamburg-Eppendorf, Hamburg
- Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No